CLINICAL TRIAL: NCT00644423
Title: Omega-3 Fatty Acids and PTSD
Brief Title: Omega-3 Fatty Acids and Post Traumatic Stress Disorder (PTSD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Durham VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VA IRB# 01210; VA IRB# 01210
Record Dates: First submitted 2008-03-20; First posted 2008-03-26 (Estimated); Results first posted 2019-08-20 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-07

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD; Cognition; Fish Oil; Omega-3 Fatty Acid
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Fatty Acids, Omega-3; Fish Oils

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Omega-3 Fatty Acid
  Interventions: Drug: Omega-3 Fatty Acid
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Omega-3 Fatty Acid — One capsule three times per day x 1 day (325mg EPA/225mg docosahexaenoic acid (DHA) tid) Two capsules three times per day x 1 day (650mg EPA/450mg DHA tid) Three capsules three times per day thereafter (975mg EPA/675mg DHA tid)
  Other Names: Fish Oil
  Arms: 1
Drug: Placebo — Matching Placebo
  Arms: 2

SUMMARY:
An increasing literature shows that omega-3 fatty acids provide numerous health benefits, including a variety of psychiatric symptoms and disorders including stress, anxiety, cognitive impairment, mood disorders (major depression and bipolar disorder) and schizophrenia. Omega-3 fatty acids may additionally represent a promising treatment strategy in patients with PTSD. Moreover, given its beneficial cardiovascular effects, adjunctive omega-3 fatty acids may also benefit the general health status of these veterans, who frequently present with a variety of comorbid medical disorders.

DETAILED DESCRIPTION:
See brief summary

ELIGIBILITY:
Inclusion Criteria:

1. Veterans 18-65 years of age, any ethnic group, either sex.
2. Ability to participate fully in the informed consent process.
3. Current diagnosis of PTSD .
4. No anticipated need to alter medications for the 10-week duration of the study.

Exclusion Criteria:

1. Serious unstable medical illness, history of traumatic brain injury (TBI) with loss of consciousness greater than 30 minutes, or history of cerebrovascular accident, prostate or breast cancer.
2. Current active suicidal and/or homicidal ideation, intent or plan.
3. Use of aspirin, warfarin or other anticoagulant therapy, as omega-3 fatty acids may increase bleeding time. Other concomitant medications for medical conditions will be addressed on a case-by-case base and determined if exclusionary.
4. Regular use of omega-3 fatty acid supplementation within the last 3 months (cod liver oil, other fish oil, flaxseed).
5. Regular consumption of more than one serving of fatty fish per week.
6. Substance dependence within the last 4 weeks (other than nicotine dependence).
7. Current Diagnostic and Statistical Manual, Fourth Edition (DSM-IV) diagnosis of bipolar disorder, schizophrenia or other psychotic disorder, or cognitive disorder due to a general medical condition other than TBI.
8. Female patients who are pregnant or breast-feeding.
9. Known allergy to study medication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-09-22 (Actual); Primary Completion 2010-07-15 (Actual); Study Completion 2010-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine E Marx, MD,MA, Principal Investigator — Durham VA Medical Center
Locations (1):
- Durham VA Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 18 participants enrolled; 11 participants started (randomized at Week 2) after a 2-week placebo lead in
Period: Overall Study
Arm/Group | Omega-3 Fatty Acid | Placebo
Started | 6 | 5
Completed | 5 | 4
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omega-3 Fatty Acid | Placebo | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 11
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.0 (10.67) | 43.6 (18.83) | 40.9 (14.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Clinician-Administered PTSD Scale (CAPS)
Description: Mean change scores in posttraumatic stress disorder symptoms (Week 10 (Week 8 Post-Randomization) minus Week 2 (Baseline)). Scores may range from 0 (no symptoms) to 136 (severe symptoms; score of 136 is based on the first 17 CAPS items administered). A reduced CAPS score indicates a reduction in (improvement) PTSD symptoms, while an increase in CAPS score indicates an increase (worsening) in PTSD symptoms.
Time Frame: Week 2 (Baseline) and Week 10 (Week 8 Post-Randomization)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Omega-3 Fatty Acid | Placebo
Number analyzed (Participants) | 6 | 5
units on a scale | -6.50 (5.124) | -18.60 (7.961)

2. Primary Outcome: Brief Assessment of Cognition in Affective Disorders (BAC-A)
Description: Mean change scores to assess cognitive changes (Week 10 (Week 8 Post-Randomization) minus Week 2 (Baseline)). The BAC-A includes brief assessments of executive functions, verbal fluency, attention, verbal memory, working memory and motor speed. Z-scores are calculated from composite scores. Higher z-scores are indicative of better cognitive performance, lower z-scores are indicative of lower cognitive performance. Range of z-scores anticipated to be between -3 and 3. Mean change scores from week 2 and week 10 (Week 2 minus Week 10).
Time Frame: Week 2 (Baseline) and Week 10 (Week 8 Post-Randomization)
Measure: Mean (Standard Error); unit: Z-score
Arm/Group | Omega-3 Fatty Acid | Placebo
Number analyzed (Participants) | 6 | 5
Z-score | 0.2583 (0.2078) | 0.2860 (0.1652)

3. Secondary Outcome: Quick Inventory of Depressive Symptomatology (QIDS)
Description: Mean change scores in depressive symptomatology (Week 10 (Week 8 Post-Randomization) minus Week 2 (Baseline)). The QIDS total scores range from 0 to 27. Total score is obtained by adding the scores for each of the nine symptom domains of the DSM-IV Major Depressive Disorder (MDD) criteria: depressed mood,loss of interest or pleasure,concentration/decision making,self-outlook,suicidal ideation, energy/fatigability, sleep,weight/appetite change, and psychomotor changes. Each item is rated 0-3 (0=least or no severity, 3=greatest severity). Higher values reflect more severe symptoms.
Time Frame: Week 2 (Baseline) and Week 10 (Week 8 Post-Randomization)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Omega-3 Fatty Acid | Placebo
Number analyzed (Participants) | 6 | 5
units on a scale | 1.167 (2.056) | -1.000 (1.000)

4. Secondary Outcome: Connor Davidson Resilience Scale (CD-RISC)
Description: Mean change scores in resiliency (Week 10 (Week 8 Post-Randomization) minus Week 2 (Baseline)). The CD-RISC was developed and tested as (i) a measure of degree of resilience, (ii) as a predictor of outcome to treatment with medication or psychotherapy, stress management and resilience-building, (iii) as a marker of progress during treatment, and (iv) as a marker of biological changes in the brain. The scale comprises 25 items, each rated on a 5-point scale (0-4) for a total range of 0-100, with higher scores reflecting greater resilience.
Time Frame: Week 2 (Baseline) and Week 10 (Week 8 Post-Randomization)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Omega-3 Fatty Acid | Placebo
Number analyzed (Participants) | 6 | 4
units on a scale | -2.000 (3.759) | 1.000 (5.986)

5. Secondary Outcome: Continuous Performance Test (CPT)
Description: Mean change scores in inpulsivity (Week 10 (Week 8 Post-Randomization) minus Week 2 (Baseline)). Computer test. Patient is to press button if target appears, but not at non-target. Impulsivity variables during test: CE=percent of response to non-target; ANT=percent of responses prior to target presentation. Results are converted to Q-scores (age and sex-adjusted normalized scores with a mean=0 and standard deviation=1 in the general population, expressing the probability determined by the Gamma function in terms of standard deviation of Gaussian density). Higher scores reflect more severe symptoms.
Time Frame: Week 2 (Baseline) and Week 10 (Week 8 Post-Randomization)
Population: Missing CPT scores from 2 participants in the Omega-3 Fatty Acid arm.
Measure: Mean (Standard Error); unit: Q-score
Arm/Group | Omega-3 Fatty Acid | Placebo
Number analyzed (Participants) | 4 | 5
Q-score | 0.6920 (0.3369) | 0.6198 (0.2911)

6. Secondary Outcome: Trail Making A
Description: Mean change scores in cognition and attention (Week 10 (Week 8 Post-Randomization) minus Week 2 (Baseline)). Trail Making Test is a measure used to assess cognition and attention. Trail Making, Part A is a timed test that consists of 25 circles on a piece of paper with the numbers 1-25 written randomly in circles. The respondent is asked to draw a line from number one, and so on, in correct numerical order, until they reach number 25. Results are reported as the number of seconds required to complete the task. Higher scores indicate greater impairment.
Time Frame: Week 2 (Baseline) and Week 10 (Week 8 Post-Randomization)
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Omega-3 Fatty Acid | Placebo
Number analyzed (Participants) | 5 | 4
seconds | -3.140 (2.112) | -11.14 (1.570)

7. Secondary Outcome: Trail Making B
Description: Mean change scores in attention and cognition (Week 10 (Week 8 Post-Randomization) minus Week 2 (Baseline)). Trail Making Test is a measure used to assess cognition and attention. Trail Making, Part B is a timed test that consists of 25 circles on a piece of paper with both numbers (1 - 13) and letters (A - L); the patient draws lines to connect the circles in an ascending pattern, but with the added task of alternating between the numbers and letters (i.e., 1-A-2-B-3-C, etc.). The respondent is asked to draw a line from number one, and so on,in correct numerical/alphabetical order, until they reach number 13. Results are reported as the number of seconds required to complete the task. Higher scores indicate greater impairment.
Time Frame: Week 2 (Baseline) and Week 10 (Week 8 Post-Randomization)
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Omega-3 Fatty Acid | Placebo
Number analyzed (Participants) | 5 | 4
seconds | -20.84 (11.77) | -30.65 (24.17)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected following the two-week placebo-lead phase and at each subsequent study visit and telephone check-in (every two weeks for 8 weeks).
Arm/Group | Omega-3 Fatty Acid | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 6/6 | 5/5
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omega-3 Fatty Acid (N=6) | Placebo (N=5)
Sweating (General disorders) | 2 (4) | 2 (2)
Drowsiness (General disorders) | 2 (3) | 2 (2)
Dry Mouth (General disorders) | 3 (4) | 1 (1)
Excitement/Agitation (General disorders) | 2 (3) | 2 (2)
Cramps (General disorders) | 1 (1) | 2 (4)
Dermatological (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (2)
Restlessness (General disorders) | 3 (5) | 0 (0)
Increased Appetite (General disorders) | 1 (2) | 2 (2)
Decreased Interest in Sex (General disorders) | 2 (2) | 1 (1)
Dizziness (General disorders) | 2 (2) | 1 (1)
Decreased Appetite (General disorders) | 1 (1) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 2 (3) | 0 (0)
Disorientation (General disorders) | 1 (1) | 1 (2)
Headache (General disorders) | 0 (0) | 2 (3)
Malaise (General disorders) | 1 (1) | 1 (2)
Nausea (General disorders) | 1 (2) | 1 (1)
Increased Motor Activity (General disorders) | 1 (1) | 1 (1)
Menstrual Disturbance (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Muscle Pain/Stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Insomnia (General disorders) | 1 (2) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (2)
Akathisia (General disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Decreased Motor Activity (General disorders) | 0 (0) | 1 (1)
Hypersomnia (General disorders) | 0 (0) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1) | 0 (0)
Impaired Sex Performance (General disorders) | 0 (0) | 1 (1)
Joint Pain/Stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nasal Congestion (General disorders) | 0 (0) | 1 (1)
Tremor (General disorders) | 0 (0) | 1 (1)
Vertigo (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes